CLINICAL TRIAL: NCT02856347
Title: Prospective Study Evaluating the Medullary Thyroid Cancer Management's Care Using PET ( Positron Emission Tomography) F-DOPA in Patients With a High Level of Postoperative Residual Thyrocalcitonin
Brief Title: Prospective Study Evaluating the Medullary Thyroid Cancer Management's Care Using PET F-DOPA in Patients With a High Level of Postoperative Residual Thyrocalcitonin
Acronym: CMTpostopFDOPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16VADS03
Record Dates: First submitted 2016-07-27; First posted 2016-08-04 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Medullary Thyroid Cancer
Keywords: Medullary Thyroid Cancer; PET F-DOPA; 18-FDOPA
MeSH Terms: conditions — Carcinoma, Medullary | interventions — fluorodopa F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET 18-FDOPA (Other): 18F-DOPA will be administered with an activity of 1.5-4 MBq/kg (MegaBecquerel) in the IV (Intra venous) tubing to decrease the extravasation risk and tracer lymphatic migration. The injection site will be distant from pathologic area (forearm).
  PET CT exam will start 10 min after tracer injection and will cover the whole body (10 to 30 min).
  Other series of images will be done 50 min after tracer injection. Images will be interpreted.
  Interventions: Other: 18F-DOPA

INTERVENTIONS:
Other: 18F-DOPA — Injection of 18F-DOPA and PET / CT-scan assessment

SUMMARY:
The aim of the trial is to study a radiating diagnosis agent used in post surgery when the biological assessment highlighted a residual disease.

This is an inter-regional multicentric, prospective study evaluating the benefit of PET F-DOPA imaging in involved node detection compared to standard imaging assessment in patient with medullary thyroid cancer.

The purpose of the study is to evaluate the impact and performance of a new PET / CT (computerized tomography ) tracer targeting dopamine receptor in patient with residual ganglionar biological disease after initial surgery of medullary thyroid cancer compared to standard imaging.

Obtained data will be compared to the "gold standard" based on :

* nodes cytology when they could be punctured
* histology when a new surgery will be recommended
* surveillance when the 2 first cases will be not applicable (imaging monitoring, evolution of thyrocalcitonin)

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18 years.
2. Patient with medullary thyroid cancer (sporadic or hereditary form).
3. Patient treated by total thyroidectomy with uni or bi-lateral lymph node dissection (in the central and/or lateral neck compartment).
4. Patient with elevated thyrocalcitonin rate > or = 150 pg/ml assessed within 6 weeks or more after surgery.
5. Patient with standard imaging assessment performed during 3 months before PET 18-FDOPA.
6. Standard imaging assessment including at least a cervical ultra-sound, a cervico-thoracic CT-scan and/or a cervico-thoraco-abdomino-pelvic CT-scan and a liver MRI.
7. Patient able to be followed at least 6 months after PET 18-FDOPA.
8. If women are breastfeeding, nursing should be discontinued during 24 hours after PET 18-FDOPA.
9. Patient must provide written informed consent prior to any specific procedure or assessment.
10. Patient must be affiliated to the French Social Security System.

Exclusion Criteria:

1. Pregnant patient.
2. Post-operative radiotherapy initiated before PET 18-FDOPA.
3. Patient with PET 18-FDG performed within 24 hours before PET 18-FDOPA.
4. Participation in any other clinical trial for therapeutic use.
5. Patient with PET / CT-scan exam contra-indication.
6. Any serious and/or unstable pre-existing psychological, familial, geographic or social condition that could interfere with medical follow-up and compliance to study procedures.
7. Patient protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Relative rate of TRUE positive nodes with PET F-DOPA compared to standard imaging assessment. | up to 3 years
  Analysis will be performed by node.

SECONDARY OUTCOMES:
Relative rate of TRUE positive nodes with PET F-DOPA compared to standard imaging assessment. | up to 3 years
  Analysis will be performed by patient.
Relative rate of FALSE positive nodes with PET F-DOPA compared to standard imaging assessment. | up to 3 years
  Analyses will be performed by patient and by node.
Relative rate of TRUE positive and FALSE metastasis with PET F-DOPA compared to standard imaging assessment. | up to 3 years
  Analyses will be performed by patient and by metastasis.
Modification rate of patient's care after PET F-DOPA exam. | up to 3 years
  Comparison of the modification of care (orientation to a surgery or a surveillance) decided after standard imaging assessment following result of TEP-FDOPA exam.
The concordance between the PET F-DOPA results of each centre and centralized review. | up to 3 years
  Concordance (centre / reviewer) of PET F-DOPA result interpretation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Slimane Zerdoud, MD, Principal Investigator — Institut Claudius Regaud
Locations (5):
- France (5):
  - CHU Haut-Lévêque, Bordeaux
  - CHU Limoges, Limoges
  - CHU Timone, Marseille
  - ICM Montpellier, Montpellier
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided